CLINICAL TRIAL: NCT04291170
Title: Comparison of Upper Extremity and Lower Extremity Function and Quick DAS
Brief Title: Comparison of Upper Extremity and Lower Extremity Function and Quick DASH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics (Research Staffing)
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 55019
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hand Injuries
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QDASH (Experimental): Completing the tasks on the QuickDASH
  Interventions: Other: QDASH
- KOOSJR (Active Comparator): Completing the tasks on the KOOSJR
  Interventions: Other: KOOSJR

INTERVENTIONS:
Other: QDASH — completing the tasks on the QDASH: open jar, wash wall, carry shopping bag, wash back, cut food, hammer wood
  Arms: QDASH
Other: KOOSJR — completing tasks on the KOOSJR: pivot, straighten, go up/down stairs, stand upright, rise from sitting, bend over
  Arms: KOOSJR

SUMMARY:
Patient reported outcome measure (PROM) are a method by which to assess outcomes from a patient perspective. The QuickDASH is a commonly used PROM. QDASH was validated against grip strength and ability work, however not against its ability to actually measure what it sets forth to measure (ie: patient's ability to use a hammer, carry a shopping bag, wash a wall, etc). The purpose of this study is to correlate the self-reported QDASH with patients' ability to perform the functions on the QDASH and compare to a control group who completes the task on a lower extremity PROM, KOOS JR.

ELIGIBILITY:
Inclusion Criteria:

* new patient
* stanford hand surgery clinic patient

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2040-09 (Estimated); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
QDASH score | Immediately after completing the taks
  the quickdash is a validated outcome measure for hand function, scored 0-100 with higher scores indicating worse disability which is bad.

CONTACTS AND LOCATIONS:
Overall Officials: Robin N Kamal, MD MBA, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD